CLINICAL TRIAL: NCT00578279
Title: Endoscopic Ultrasound-guided Celiac Plexus Neurolysis (EUS-CPN) With Alcohol in Patients With Locally Advanced and Unresectable Pancreatic Adenocarcinoma: A Randomized Pilot Study
Brief Title: Endoscopic Ultrasound-guided Celiac Plexus Neurolysis (EUS-CPN)With Alcohol in Unresectable Pancreatic Cancer: a Pilot Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0702-25; IRB # 0702-25; Clarian Values Grant: vfr-262
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Results first posted 2012-10-19 (Estimated); Last update posted 2012-10-19 (Estimated); Status verified 2010-06

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Other): subject randomized to 10ml of dehydrated alcohol
  Interventions: Drug: dehydrated alcohol
- B (Experimental): subject randomized to 20ml of dehydrated alcohol
  Interventions: Drug: dehydrated alcohol

INTERVENTIONS:
Drug: dehydrated alcohol — subject randomized to 10ml or 20ml of dehydrated alcohol one time during the EUS-CPN procedure

SUMMARY:
The purpose of this study is to obtain preliminary safety and efficacy data after endoscopic ultrasound-guided celiac plexus neurolysis (EUS-CPN) in patients with locally advanced or unresectable pancreatic adenocarcinoma.

Hypotheses:

1. Increased amounts of alcohol used in EUS-CPN is safe and more efficacious in improving pain relief in patients with locally advanced or unresectable pancreatic adenocarcinoma.
2. Effective pain relief obtained from EUS-CPN will be related to better quality of life (QOL)

ELIGIBILITY:
Inclusion Criteria:

* A total of 20 consecutive subjects with locally advanced or unresectable pancreatic adenocarcinoma (stage II to IV) with pain (abdominal and/or back). Subjects with known or suspected unresectable pancreatic adenocarcinoma will be recruited for this study, as a diagnosis of unresectable pancreatic adenocarcinoma is often made during the endoscopic ultrasound (EUS) procedure.
* Subjects must have documented disease by computed tomography (CT), endoscopic retrograde cholangio-pancreatography (ERCP), or EUS.
* Subjects undergoing EUS for pancreatic cancer staging.
* Subjects undergoing pancreatic cancer surgery are eligible for study entry beginning 5 days after the operation if they have not had an intraoperative celiac plexus neurolysis.
* No evidence of dementia or altered mental status that would prohibit the giving and understanding of informed consent, and no evidence of psychiatric risk that would preclude adequate compliance with this protocol.

Subjects must not have a coagulopathy (platelet <50,000, INR>1.5, or bleeding disorder, or on blood thinners) Subjects with platelets below 50,000 will not be eligible to participate in this study due to the risk of bleeding. Patients will be asked to discontinue use of non-steroidals for 5 days prior to the procedure. Patients on plavix will be asked to discontinue use for 7 days prior to the procedure if they are clinically able to do so. Patients on coumadin or lovenox will also need to discontinue use prior to the procedure, but decisions regarding their management will be made on an individual basis as per our usual standards of care.

* Subjects must provide signed written informed consent.
* A baseline pain score is not required, however, subjects must be having pain that is requiring a stable dose of pain medication for control of pain.

Exclusion Criteria:

* Subjects will be excluded if they have undergone a celiac plexus neurolysis (endoscopic, percutaneous, or surgical).
* Presence of an implanted epidural or intrathecal analgesic therapy. Subjects with psychiatric illness that affects their ability to assess quality of life or compliance with the protocol.
* Subjects with uncorrectable coagulopathy
* Subjects with an allergy to bupivacaine or alcohol.
* Presence of an aneurysm in the abdominal aorta, celiac trunk, or superior mesenteric artery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julia LeBlanc, MD, MPH, Principal Investigator — Indiana University
Locations (1):
- Clarian Health: Indiana University Hospital, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 10 mL of Alcohol Injection: subject randomized to 10ml of dehydrated alcohol
- 20 mL of Alcohol Injection: subject randomized to 20ml of dehydrated alcohol
Period: Overall Study
Arm/Group | 10 mL of Alcohol Injection | 20 mL of Alcohol Injection
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 10 mL of Alcohol Injection | 20 mL of Alcohol Injection | Total
Number analyzed (Participants) | 10 | 10 | 20
Age Continuous [Mean (Standard Deviation); unit: years] | 66 (14) | 63 (10) | 64 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 5 | 4 | 9
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: The Change in Mean Pain Scale Rating in Patients Following Treatment With 10mL or 20mL of Alcohol Injection
Description: Pain will be assessed at baseline 24 hours after the procedure and weekly thereafter, until the subject reports no subjective pain relief from the procedure. Pain relief is defined as a decrease in 2 points on a 0-10 point pain rating scale. Zero is no pain and 10 is the worst pain.
Time Frame: baseline up to 1 year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 10 mL of Alcohol Injection | 20 mL of Alcohol Injection
Number analyzed (Participants) | 10 | 10
units on a scale | 7.9 (10.8) | 8.4 (9.2)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | 10 mL of Alcohol Injection | 20 mL of Alcohol Injection
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No